CLINICAL TRIAL: NCT04939792
Title: Optimization of Blood Levels of 25(OH)-Vitamin D in African Americans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Sushil Jain, Principle Investigator, Louisiana State University Health Sciences Center Shreveport
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRP-503
Record Dates: First submitted 2021-06-08; First posted 2021-06-25 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Vitamin D Deficiency
Keywords: African American;; Vitamin D;; Insulin resistance; Alzheimer's Disease
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Alzheimer Disease | interventions — Vitamin D; Cholecalciferol; Starch; Cysteine; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Initially, all of the study subjects will be provided placebo supplementation as a placebo run-in period for one month before randomization. The placebo run-in period is meant to stabilize subjects in the study and will prevent any effect due solely to inclusion in the study. Placebo and supplement capsules will be similar in appearance, taste, texture, and smell, and will be provided by the pharmacist, who will have the codes for which subjects are assigned to which supplement or placebo.
  During testing, the placebo group will take two placebo capsules a day in the morning. Supplements will be taken daily with food at breakfast for 6 months, while participants continue to carry on a normal lifestyle
  Interventions: Drug: Placebo
- L-Cysteine (Experimental): LC group will receive two capsules of LC daily. Supplements will be taken daily with food at breakfast for 6 months, while participants continue to carry on a normal lifestyle
  Interventions: Drug: L-cysteine
- Vitamin D3 (Experimental): VD group will take two capsules and each capsule will contain 1000 IU VD daily. Supplements will be taken daily with food at breakfast for 6 months, while participants continue to carry on a normal lifestyle
  Interventions: Drug: Vitamin D
- Vitamin D3 and L-Cysteine (Experimental): VD+LC group will take daily two capsule containing 1000 IU+500 mg LC. Supplements will be taken daily with food at breakfast for 6 months, while participants continue to carry on a normal lifestyle
  Interventions: Drug: Vitamin D + L-cysteine

INTERVENTIONS:
Drug: Vitamin D — Capsules ingested orally
  Other Names: cholecalciferol
  Arms: Vitamin D3
Drug: Placebo — Capsule ingested orally
  Other Names: starch
  Arms: Placebo
Drug: Vitamin D + L-cysteine — Capsule ingested orally
  Other Names: combination of vitamin D and L-cysteine
  Arms: Vitamin D3 and L-Cysteine
Drug: L-cysteine — Capsule ingested orally
  Other Names: amino acid
  Arms: L-Cysteine

SUMMARY:
Two-thirds of the US population, particularly African Americans (AA), is at risk for inadequate or deficient 25-hydroxy-vitamin D (25(OH)VD). Epidemiological studies demonstrate an association between better health outcomes and higher blood levels of 25(OH)VD . Randomized controlled clinical trials have shown that, while supraphysiological high doses of VD are needed to achieve adequate blood levels of 25(OH)VD, not all subjects respond to them. Recent studies have also questioned the therapeutic effects of high-dose VD supplementation. Severe VD deficiency has been associated independently with the future risk of mild cognitive impairment (MCI) and dementia. A reduction in GSH and an increase in the oxidative stress levels of serum, erythrocytes, and circulating lymphocytes has been observed in MCI and Alzheimer disease, findings similar to those in VD deficient persons. Scholarly reviews conclude that excess oxidative stress is one of the major risk factors for AD and support a potential therapeutic role for L-cysteine (LC, a GSH precursor) and vitamin D (VD) supplementation in the treatment of Alzheimer disease symptoms. This application presents the investigators' design for a randomized, double-blind, placebo-controlled clinical trial to test the hypothesis that supplementation with VD in combination with L-cysteine (LC) is more successful at optimizing the statuses of 25(OH)VD [biological signatures] and simultaneously decreasing TNF-α, IR [functional or clinical outcomes], and oxidative stress, suggesting a better therapeutic approach compared with supplementation with VD alone in AA subjects.

ELIGIBILITY:
Inclusion Criteria:

* African American volunteers only
* Participants between the ages of 18 and 65
* Must be In good general health
* Women with negative pregnancy tests

Exclusion Criteria:

* Subjects with Diabetes, Heart disease, Sickle Cell disease, or Epilepsy
* Subjects with serum positive pregnancy test or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
25-hydroxy-vitamin D | 6 months
  Change in blood levels of 25(OH)VD

SECONDARY OUTCOMES:
TNF-α | 6 months
  Whether any increase in vitamin D beneficially decreases insulin resistance
HOMA-IR | 6 months
  Whether any decrease in TNF-a beneficially decreases insulin resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Louisiana State University Health Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study
Supporting Information: Study Protocol, CSR
Time Frame: 3 years

REFERENCES:
- [Derived] Jain SK, Justin Margret J, Zachary A Jr, Lally MM, Vanchiere JA, Mhanna MJ, Shi R, Levine SN. Effects of vitamin D and L-cysteine cosupplementation on circulating bioavailable and total 25-hydroxy-vitamin D, the free/total testosterone ratio and inflammatory biomarkers in healthy vitamin D-deficient African Americans: a placebo-controlled double-blind clinical trial. BMJ Nutr Prev Health. 2024 Aug 7;7(2):e000856. doi: 10.1136/bmjnph-2023-000856. eCollection 2024. PMID 39882299

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT04939792/Prot_000.pdf
  • Informed Consent Form (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT04939792/ICF_001.pdf